CLINICAL TRIAL: NCT05743582
Title: Analysis of Innate Immune Competence in People With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Innate Immunity in COPD
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC23003
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Alveolar macrophages; Peripheral blood mononuclear cells; Neutrophils; Bactericidal mechanisms; Immune cell metabolism; Epigenetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy; Specimen Handling; Blood Donation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Immune cells from bronchoalveolar lavage obtained by bronchoscopy and peripheral blood mononuclear cells/neutrophils obtained from peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD patients: Bronchoscopy to retrieve bronchoalveolar lavage fluid for isolation of immune cells, and phlebotomy for blood sample collection.
  Interventions: Procedure: Bronchoscopy for sample collection; Procedure: Blood donation
- Healthy controls - smokers: Bronchoscopy to retrieve bronchoalveolar lavage fluid for isolation of immune cells, and phlebotomy for blood sample collection.
  Interventions: Procedure: Bronchoscopy for sample collection; Procedure: Blood donation
- Healthy controls - non-smokers: Bronchoscopy to retrieve bronchoalveolar lavage fluid for isolation of immune cells, and phlebotomy for blood sample collection.
  Interventions: Procedure: Bronchoscopy for sample collection; Procedure: Blood donation

INTERVENTIONS:
Procedure: Bronchoscopy for sample collection — Participants will undergo a single bronchoscopy and bronchoalveolar lavage to obtain immune cells.
Procedure: Blood donation — Participants will donate a single blood sample for isolation of immune cells from peripheral blood.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) causes obstruction to airflow when breathing out. It is a leading cause of chronic lung disease, hospitalization and death. Smoking is the major cause of COPD but why some smokers develop COPD while others do not is poorly understood. A central feature of COPD is accumulation of inflammatory blood cells, macrophages and neutrophils, in the airway, leading to lung injury and airway damage. The small airways of many patients with COPD contain bacteria, which are absent in healthy smokers or non-smokers. These bacteria stimulate recruitment of neutrophils, macrophages and other inflammatory cells, further accelerating airway injury. The investigators and others have shown resident macrophages in the lung and inflammatory cells (neutrophils and macrophages) recruited from the blood, which normally clear bacteria, have reduced anti-bacterial capacity in COPD and that their altered function impairs the resolution of inflammation. The investigators now wish to test why these cells fail to clear bacteria focusing in particular on how they use molecules as food to generate energy, a process termed metabolism, since this is an important determinant of immune cell function. Comparison will be made between lung resident cells (obtained by performing bronchoscopy and washing a segment of lung to flush out immune cells) and those from the blood to determine if the alterations are specific to the lung. The investigators will identify alterations in responses to bacteria in relation to changes in metabolism . A major focus will be on how structures in the cell that normally are key for energy production (i.e. mitochondria) become dysfunctional and how this impacts responses to bacteria. The investigators will relate findings to the clinical features of COPD and to healthy non-smokers and smokers to separate smoking-related changes from COPD. The aim is to develop new approaches with which to treat and manage COPD.

DETAILED DESCRIPTION:
COPD has become one of the major causes of ill health throughout the world. COPD has major economic impact being the second commonest causes of hospital admission and days lost to work in the UK where an estimated 10% of the population over 40 are affected. The disease causing mechanisms are not well defined but a central feature is development of a chronic inflammatory process. Inflammation in COPD is progressive and persists after inciting factors, such as cigarette smoke, are removed. The stimuli to persistent inflammation and the failure of normal cues to resolve this inflammation are poorly characterised. Lung inflammation in COPD is largely resistant to the antiinflammatory actions of corticosteroids, currently used as treatment, which fail to modify disease progression or mortality. Existing therapeutic approaches for COPD are therefore flawed and do not alter the central chronic inflammatory process.

Better understanding of COPD pathogenesis is essential if new therapeutic strategies are to be developed that will alter the course of the disease. A sub-set of COPD patients have more frequent exacerbations, which are associated with more rapid decline in pulmonary function tests and increased mortality. Bacterial infection is a frequent cause of these exacerbations. In addition some of the high-risk patients with COPD are more susceptible to bacterial pneumonia. In COPD, the lower respiratory tract is colonised with a higher density of bacteria (including Haemophilus influenzae or Streptococcus pneumoniae), whereas in non-smoking subjects and smokers with normal lung function the density of bacteria is much lower. This suggests there may be a defect in immune responses to bacteria in patients with COPD, in particular involving the part of the immune response which is termed 'innate', which provides the most rapid and generic response to bacteria.

Lung host defence against bacteria requires the co-ordinated action of both immune cells and factors released into the airway termed humoral factors. Alveolar macrophage (AM) competence is essential to maintain sterility in the lower airway and bacterial phagocytosis and killing is complemented by a delayed programme of cell death termed apoptosis, which provides a significant increment to bacterial killing and shuts off the inflammatory response. When this component of host defence is over-whelmed recruited cells that ingest bacteria termed phagocytes (i.e. neutrophils and macrophages) become key effectors of the host response. Research suggests that monocyte-derived macrophages (MDM) isolated from patients with COPD have impaired capacity for phagocytosis of bacteria as compared to healthy donors or smokers without COPD. That this defect is apparent in cells isolated from the blood suggests it may reflect a systemic defect in bacterial clearance. In addition there is a marked defect in AM isolated from the lung, suggesting additional defects imposed by the lung environment, that impacts uptake of bacteria coated with antibody. The investigators have also shown that macrophages are impaired in their ability to kill the bacteria they ingest. The molecular basis of the decreased clearance of bacteria is unclear but research by the investigators has found that macrophages fail to produce an increment in a factor that kills bacteria that is produced by mitochondria, termed mitochondrial reactive oxygen species (mROS) and this may contribute to both impaired ingestion and killing of bacteria.

Mitochondria are structures in cell that generate energy but how they burn fuels in the form of molecules adapts to aid immune function. The investigators believe that in COPD mitochondria in macrophages fail to adapt during bacterial challenge and this underpins the immune defect observed for bacteria. Similarly, the investigators have shown that peripheral blood neutrophils have impaired killing of bacteria in COPD and that this is associated with impaired gluconeogenesis, a process that stores glucose in the form of glycogen. This glycogen is normally used by neutrophils as a source of glucose to help prime responses to bacteria and this defect in COPD neutrophils impairs their capacity to kill bacteria This has not been previously addressed and the investigators will focus on four main aspects: i) the molecules myeloid cells burn as fuel sources during metabolism in COPD in at rest and in response to bacteria and other inflammatory stimuli, ii) alterations in mitochondrial function in myeloid cells in COPD, iii) whether alterations are confined to myeloid cells in the lung or expressed at sites removed from the lung and the mechanisms of these effects and iv) methods to recalibrate altered responses determined by the investigators in myeloid cells in COPD. The cells and materials that will be generated will allow additional research and will be used to help test other hypotheses and identify additional mechanism underlying immune dysfunction and promotion of inflammation in COPD that emerge as work by the investigators and the field progresses during the lifetime of this research.

ELIGIBILITY:
Inclusion Criteria:

COPD patients:

* COPD patients aged 18-77 years who are GOLD Stage 1 or 2 or 3; for patients undergoing bronchoscopy already for a clinical reason.
* COPD patients aged 18-77 years old who are GOLD Stage 1,2 or 3 for patients who are donating blood only.
* COPD patients aged 18-69 years who are GOLD Stage 1 or 2 for patients undergoing bronchoscopy for research purposes.
* COPD- Defined by radiological investigation of chest either chest X-ray or High-resolution CT scan in previous 12 months
* Ability to provide informed consent

Healthy volunteers:

* Any healthy volunteer aged 18-77 years
* Ability to provide informed consent

Exclusion Criteria:

COPD patients:

* Individuals known to have active malignancy, immunosuppression, diabetes mellitus, chronic kidney disease or hepatic failure.
* Individuals with a history of anaemia
* Individuals who have donated >250 ml of blood for any reason within the last 6 months
* Individuals who are pregnant or breast feeding.
* Current participation in any other clinical trial, except those directly relating to this cohort and study.
* Individuals who have had a febrile illness or other symptoms of acute infectious illness (respiratory, enteric or soft tissue) within the last 2 weeks
* Individuals who have received a vaccine in the past 2 weeks
* Inability to communicate in English or convey willingness to participate.
* For bronchoscopy - Any significant lung condition that would contra-indicate bronchoscopy including:

active acute lung infection (with the exception of asymptomatic pulmonary colonisation) or malignancy, significant coexisting interstitial lung disease or additional pulmonary diagnosis in addition to COPD.

Healthy volunteers:

* Individuals known to have active malignancy, immunosuppression, diabetes mellitus, chronic kidney disease or hepatic failure
* Individuals with anaemia on the screening full blood count (FBC)
* Individuals who donated >250 ml of blood for any reason within the last 6 months
* Individuals who are pregnant or breast feeding
* Current participation in any other clinical trial
* Individuals who have had a febrile illness or other symptoms of acute infectious illness (respiratory, enteric or soft tissue) within the last 2 weeks.
* Individuals who have received a vaccine in the past 2 weeks
* Chronic or acute respiratory disease.
* Any chronic medical condition or receipt of regular prescription medication other than the oral contraceptive pill.
* Inability to communicate in English or convey willingness to participate
* For bronchoscopy - Any active lung condition including any lung infection or asthma Any significant abnormality on CXR that would contraindicate bronchoscopy FEV1 <65% predicted (BTS Guidelines, 2001)

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 189 participants split evenly into: COPD patients, healthy smokers, healthy non-smokers (63 each)
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Identification of immunometabolic responses in immune cells required for microbicidal activity. | 5 years
  This programme will identify core features of the immunometabolic response and of mitochondrial function that are required for optimal macrophage responses to bacteria and establish how these core responses are perturbed in COPD. Outcomes will be related back to clinical phenotypes of the patients enrolled in the study. The investigators will also develop models and therapeutic approaches with which to translate this programme and suggest approaches for future clinical trials that may include use of repurposed agents.

CONTACTS AND LOCATIONS:
Overall Officials: David H Dockrell, MD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - University of Edinburgh, Edinburgh
  - Royal Infirmary of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared, in anonymised form only, upon request. No identifiable personal information will be used when publishing results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will become available upon publication of results at the end of the study.
Access Criteria: IPD will be shared directly with other researchers for analysis of cohort data upon request from the Principal Investigator.

REFERENCES:
- [Background] Dockrell DH, Marriott HM, Prince LR, Ridger VC, Ince PG, Hellewell PG, Whyte MK. Alveolar macrophage apoptosis contributes to pneumococcal clearance in a resolving model of pulmonary infection. J Immunol. 2003 Nov 15;171(10):5380-8. doi: 10.4049/jimmunol.171.10.5380. PMID 14607941
- [Background] Taylor AE, Finney-Hayward TK, Quint JK, Thomas CM, Tudhope SJ, Wedzicha JA, Barnes PJ, Donnelly LE. Defective macrophage phagocytosis of bacteria in COPD. Eur Respir J. 2010 May;35(5):1039-47. doi: 10.1183/09031936.00036709. Epub 2009 Nov 6. PMID 19897561
- [Background] Bewley MA, Preston JA, Mohasin M, Marriott HM, Budd RC, Swales J, Collini P, Greaves DR, Craig RW, Brightling CE, Donnelly LE, Barnes PJ, Singh D, Shapiro SD, Whyte MKB, Dockrell DH. Impaired Mitochondrial Microbicidal Responses in Chronic Obstructive Pulmonary Disease Macrophages. Am J Respir Crit Care Med. 2017 Oct 1;196(7):845-855. doi: 10.1164/rccm.201608-1714OC. PMID 28557543
- [Background] Bewley MA, Budd RC, Ryan E, Cole J, Collini P, Marshall J, Kolsum U, Beech G, Emes RD, Tcherniaeva I, Berbers GAM, Walmsley SR, Donaldson G, Wedzicha JA, Kilty I, Rumsey W, Sanchez Y, Brightling CE, Donnelly LE, Barnes PJ, Singh D, Whyte MKB, Dockrell DH; COPDMAP. Opsonic Phagocytosis in Chronic Obstructive Pulmonary Disease Is Enhanced by Nrf2 Agonists. Am J Respir Crit Care Med. 2018 Sep 15;198(6):739-750. doi: 10.1164/rccm.201705-0903OC. PMID 29547002
- [Background] Belchamber KBR, Singh R, Batista CM, Whyte MK, Dockrell DH, Kilty I, Robinson MJ, Wedzicha JA, Barnes PJ, Donnelly LE; COPD-MAP consortium. Defective bacterial phagocytosis is associated with dysfunctional mitochondria in COPD macrophages. Eur Respir J. 2019 Oct 10;54(4):1802244. doi: 10.1183/13993003.02244-2018. Print 2019 Oct. PMID 31320451
- [Background] Mills EL, Kelly B, O'Neill LAJ. Mitochondria are the powerhouses of immunity. Nat Immunol. 2017 Apr 18;18(5):488-498. doi: 10.1038/ni.3704. PMID 28418387
- [Background] Sadiku P, Willson JA, Ryan EM, Sammut D, Coelho P, Watts ER, Grecian R, Young JM, Bewley M, Arienti S, Mirchandani AS, Sanchez Garcia MA, Morrison T, Zhang A, Reyes L, Griessler T, Jheeta P, Paterson GG, Graham CJ, Thomson JP, Baillie K, Thompson AAR, Morgan JM, Acosta-Sanchez A, Darde VM, Duran J, Guinovart JJ, Rodriguez-Blanco G, Von Kriegsheim A, Meehan RR, Mazzone M, Dockrell DH, Ghesquiere B, Carmeliet P, Whyte MKB, Walmsley SR. Neutrophils Fuel Effective Immune Responses through Gluconeogenesis and Glycogenesis. Cell Metab. 2021 Feb 2;33(2):411-423.e4. doi: 10.1016/j.cmet.2020.11.016. Epub 2020 Dec 10. PMID 33306983